CLINICAL TRIAL: NCT03659396
Title: the Effects of Individualized Tai Chi Training on Balance Control in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Wen-Hsu Sung, Associate Professor, National Yang-Ming University, Department of Physical Therapy and Assistive Technology, National Yang Ming Chiao Tung University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000087
Record Dates: First submitted 2017-03-28; First posted 2018-09-06 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- individualized Tai Chi (Experimental): patient received individualized Tai Chi program training.
  Interventions: Other: individualized Tai Chi
- Entire Tai Chi (Active Comparator): patient received Entire Tai Chi program training.
  Interventions: Other: Entire Tai Chi
- home-based program (Placebo Comparator): patient received home-based program training.
  Interventions: Other: home-based program

INTERVENTIONS:
Other: individualized Tai Chi — individualized Tai Chi training exercise
  Arms: individualized Tai Chi
Other: Entire Tai Chi — the classical Yang style Tai Chi program
  Arms: Entire Tai Chi
Other: home-based program — Home-based exercise
  Arms: home-based program

SUMMARY:
Traditional Tai Chi is too complex for most elderly individuals. There have been few reports regarding the development of simplified Tai Chi programs to suit the physical needs of elderly adults. However, these programs were not individualized according to the participants' balance control abilities.The investigators already developed an individualized Tai Chi program. This objective of the study was to investigate the effect of individualized Tai Chi training.

DETAILED DESCRIPTION:
Background: Balance control is an important skill for human to maintain a myriad of postures and activities. The elderly suffering from balance impairment by aging have high rate to increase fall-related injuries, restricted activities, declined physical functions, and decrease quality of life. Tai Chi (TC) has been demonstrated as an innovative way to promote balance function, which is a suitable exercise for older people because of its slow movement, changeable base of supports, multi-directions weight shifting and less impact on lower extremities. Recent systematic reviews have shown that TC exercises have significant benefits in improving balance control, but most of them are only connected with healthy elderlies. Actually, the long standing time and training duration, challenged recollection by its sequence forms, and complex coordination for upper and lower extremities of TC usually make it difficult to practice for some elderlies with poor physical functions. Therefore, the method of individualized TC exercise program, integrated with biomechanical analyses, is developed in this research. It can afford an easier and more applicable training for elderly to improve the balance abilities.

Purposes:To evaluate the effects of individualized Tai Chi training on balance control in elderly.

Methods: This research is a quasi-experimental design and prospective study. Participants were recruited and assigned into individualized TC, entire TC group and home-based education group

ELIGIBILITY:
Inclusion Criteria:

Participants in the study were community-dwelling volunteers aged over 65 years. Participants were ambulatory and did not

Exclusion Criteria:

have any history of

1. diagnosed central nervous system
2. vestibular pathology
3. cognitive impairment
4. visual deficit
5. fracture of lower limb in recent 6 months
6. with Tai Chi practice experience for more than 2 months.
7. severe hearing impairment to follow instruction

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Time Up and Go | 8 weeks
  is a simple test used to assess a person's mobility and requires both static and dynamic balance

SECONDARY OUTCOMES:
Berg balance scale | 8 weeks
  The Berg Balance Scale (BBS) was developed to measure balance among older people with impairment in balance function by assessing the performance of functional tasks. 1 The scale consists of 14 items, scored from 0 to 4, which are added to make a total score between 0 and 56; a higher score indicates better balance.
functional reach | 8 weeks
  The Functional Reach Test is a quick and simple, single-task dynamic test that defines functional reach as. "the maximal distance one can reach forward beyond arm's length, while maintaining a fixed base of support in the standing position"
muscle strength of hip flexor and extensor | 8 weeks
  muscle strength of hip flexor and extensor by dynamometer
muscle strength of hip abductor and adductor | 8 weeks
  muscle strength of hip abductor and adductor by dynamometer
muscle strength of knee flexor and extensor | 8 weeks
  muscle strength of knee flexor and extensor by dynamometer
muscle strength of ankle dorsiflexor and plantarflexor | 8 weeks
  muscle strength of ankle dorsiflexor and plantarflexor by dynamometer

REFERENCES:
- [Derived] Penn IW, Sung WH, Lin CH, Chuang E, Chuang TY, Lin PH. Effects of individualized Tai-Chi on balance and lower-limb strength in older adults. BMC Geriatr. 2019 Aug 27;19(1):235. doi: 10.1186/s12877-019-1250-8. PMID 31455225